CLINICAL TRIAL: NCT00247715
Title: Comparison of an Antacid/H2-Receptor Antagonist/Proton Pump Inhibitor Versus a Proton Pump Inhibitor/H2-Receptor Antagonist/Antacid Treatment Strategy for Patients With New Onset Dyspepsia in General Practice (The DIAMOND-Study)
Brief Title: Comparison of a "Step-Up" Versus a "Step-Down" Treatment Strategy for Patients With New Onset Dyspepsia in General Practice (The DIAMOND-Study)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 945-03-052; CMO 2002/141
Record Dates: First submitted 2005-11-01; First posted 2005-11-02 (Estimated); Last update posted 2007-08-29 (Estimated); Status verified 2007-08

CONDITIONS: Dyspepsia; Gastrointestinal Diseases
Keywords: uninvestigated dyspepsia; cost effectiveness; acid suppressive medicine; primary care; gastrointestinal complaints; Gastrointestinal drugs
MeSH Terms: conditions — Dyspepsia; Gastrointestinal Diseases | interventions — Aluminum Hydroxide; Magnesium Oxide; Ranitidine; Pantoprazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Step-up (Other): Stepwise treatment:
  * step1: antacid (+placebo proton pump inhibitor)
  * step2: H2-receptor antagonist
  * step3: proton pump inhibitor (+ placebo antacid)
  Interventions: Drug: algeldrate/magnesium oxide; Drug: ranitidine; Drug: pantoprazole
- step-down (Other): Stepwise treatment:
  * step1: proton pump inhibitor (+placebo antacid)
  * step2: H2-receptor antagonist
  * step3: antacid (+proton pump inhibitor)
  Interventions: Drug: algeldrate/magnesium oxide; Drug: ranitidine; Drug: pantoprazole

INTERVENTIONS:
Drug: algeldrate/magnesium oxide
Drug: ranitidine
Drug: pantoprazole

SUMMARY:
The purpose of this study was to determine which treatment strategy, the step-up or the step-down treatment strategy, is the most cost-effective treatment for patients with new onset dyspepsia in primary care.

DETAILED DESCRIPTION:
Dyspepsia is very common in the population. On an annual basis, 20%-40% of the general population suffers from upper gastrointestinal symptoms. The prevalence of dyspepsia presenting in primary care is about 3%, on average 24% of these patients are referred for secondary care in the same year. In spite of consensus statements and guidelines, the most effective treatment strategy for managing dyspepsia in primary care remains to be determined. In 2000 the Health Council of the Netherlands published some advice for the Minister of Health, Welfare and Sport with special consideration to the most cost-effective strategies for the management of dyspepsia. The Health Counsel Committee agrees in general with the existing guidelines of the Dutch College of General Practitioners to start with empirical treatment. However, the committee concluded that more research is necessary for management of dyspepsia in primary care, especially in uninvestigated patients as most research has been conducted in patients with persistent dyspeptic symptoms referred for secondary care.

Comparison: In this study empirical treatment according to the existing guidelines of the Dutch College of General Practitioners (the step-up treatment strategy) is compared to a step-down treatment strategy. According to this step-down treatment strategy the patient begins treatment with a proton pomp inhibitor, which is an expensive acid-suppressor and is often prescribed by general practitioners.

Step-up strategy: Algeldrate-magnesium oxide, in case of persisting/relapsing symptoms continued with ranitidine, if necessary continued with pantoprazole.

Step-down strategy: Pantoprazole, in case of persisting or relapsing symptoms continued with ranitidine, if necessary continued with algeldrate-magnesium oxide.

ELIGIBILITY:
Inclusion Criteria:

* Presence of a new episode of dyspepsia, defined as episodic or persistent symptoms including abdominal pain or discomfort and which are, in the opinion of the general practitioner, referable to the upper gastrointestinal tract.
* Over 18 years of age
* Informed consent (written) given.

Exclusion Criteria:

* Use of prescribed acid suppressive medication during 3 months before consult
* Investigated by upper gastrointestinal endoscopy one year before inclusion
* Malignancy
* Contraindication to the study medication
* Pregnancy
* Alarming symptoms like weight loss, bleeding, and disturbed food passage
* Patients with insufficient comprehension of the Dutch language

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 664 (Actual)
Dates: Start 2003-10; Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Cost-efficacy | 6 months

SECONDARY OUTCOMES:
Severity of gastrointestinal symptoms | 2 weeks, after each treatment steps, and 6 months
Quality of life | 2 weeks, after each treatment step, and 6 months
Genetic and psychosocial determinants | baseline and 6 months
Patient compliance after treatment | 0 to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jan BMJ Jansen, MD, PhD, Study Chair — Radboud University Nijmegen Medical Center; Robert JF Laheij, PhD, Principal Investigator — Radboud University Nijmegen Medical Center; Niek De Wit, MD, PhD, Study Chair — UMC Utrecht; Mattijs E Numans, MD, PhD, Study Chair — UMC Utrecht; Melvin Samsom, MD, PhD, Study Chair — UMC Utrecht; Jean WM Muris, MD, PhD, Study Chair — Maastricht University; Andre Knottnerus, MD, PhD, Study Chair — Maastricht University
Locations (3):
- Netherlands (3):
  - Radboud University Nijmegen Medical Center, Nijmegen, Gelderland
  - Maastricht University, Maastricht, Limburg
  - UMC Utrecht, Utrecht, Utrecht

REFERENCES:
- [Background] Fransen GA, van Marrewijk CJ, Mujakovic S, Muris JW, Laheij RJ, Numans ME, de Wit NJ, Samsom M, Jansen JB, Knottnerus JA. Pragmatic trials in primary care. Methodological challenges and solutions demonstrated by the DIAMOND-study. BMC Med Res Methodol. 2007 Apr 23;7:16. doi: 10.1186/1471-2288-7-16. PMID 17451599
- [Derived] van Marrewijk CJ, Mujakovic S, Fransen GA, Numans ME, de Wit NJ, Muris JW, van Oijen MG, Jansen JB, Grobbee DE, Knottnerus JA, Laheij RJ. Effect and cost-effectiveness of step-up versus step-down treatment with antacids, H2-receptor antagonists, and proton pump inhibitors in patients with new onset dyspepsia (DIAMOND study): a primary-care-based randomised controlled trial. Lancet. 2009 Jan 17;373(9659):215-25. doi: 10.1016/S0140-6736(09)60070-2. PMID 19150702